CLINICAL TRIAL: NCT04345718
Title: Exemplar Hospital Initiation Trial to Enhance Treatment Engagement - Comparative Effectiveness Trial of Extended Release Buprenorphine Versus Treatment as Usual for Hospitalized Patients With Opioid Use Disorder
Brief Title: EXHIT ENTRE Comparative Effectiveness Trial
Acronym: EXHITENTRE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gavin Bart (Other)
Collaborators: Hennepin Healthcare Research Institute (Other); National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor-Investigator, Gavin Bart, Gavin Bart, MD PhD FACP DFASAM, Hennepin Healthcare Research Institute
Organization: Hennepin Healthcare Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA CTN 0098A; 5UG1DA040316-05 (NIH)
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Substance Use Disorder; Opioid Use Disorder, Moderate; Opioid Use Disorder, Severe
Keywords: MOUD; XR-BUP; ACS; OUD; SUD
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders; Lymphoma, Follicular | interventions — Dosage Forms; Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a multi-site open-label randomized comparative effectiveness trial of a 28-day formulation of XR-BUP versus TAU for hospitalized patients with OUD agreeing to MOUD. Approximately 4-5 sites (hospitals) with existing ACSs experienced in hospital-initiated MOUD will be selected. Identification of patients with OUD will occur as per each site's local practice. Approximately 314 hospitalized patients with OUD who were not receiving prescribed MOUD for at least 14 days prior to hospitalization and are willing to start MOUD including buprenorphine will be randomized 1:1 to two different strategies. After baseline assessments are performed, eligible participants will be randomized in a 1:1 ratio to XR-BUP or TAU
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Single subcutaneous injection of a 28-day formulation of extended-release buprenorphine within 72 hours of anticipated hospital discharge.
  Interventions: Drug: Extended Release Buprenorphine
- Treatment as Usual (Active Comparator): Community standard of care that includes initiation of either methadone, sublingual (SL) buprenorphine, or naltrexone prior to hospital discharge.
  Interventions: Drug: Treatment as Usual

INTERVENTIONS:
Drug: Extended Release Buprenorphine — XR-BUP administration prior to hospital discharge will increase engagement in OUD care on the 34th day following hospital discharge more than is currently afforded by ACS TAU approaches (e.g., methadone, SL-BUP, and naltrexone).
  Other Names: Medication for Opioid Use Disorder
  Arms: Interventional
Drug: Treatment as Usual — Community standard medication for opioid use disorder (e.g., methadone, sublingual buprenorphine, naltrexone) initiated prior to hospital discharge.
  Other Names: Standard Medication for Opioid Use Disorder
  Arms: Treatment as Usual

SUMMARY:
This study is a multi-site open-label randomized comparative effectiveness trial of a 28-day formulation of extended-release buprenorphine (XR-BUP) versus treatment as usual (TAU) for hospitalized patients with a moderate or severe opioid use disorder (OUD) seen by an addiction consultation service (ACS) and agreeing to initiate a medication for OUD (MOUD). Participants will be randomly assigned to XR-BUP or TAU to be received within 72 hours of anticipated hospital discharge. Follow up will occur at approximately 34, 90, and 180 days following hospital discharge.

DETAILED DESCRIPTION:
The study will randomize approximately 314 hospitalized men and women ages 18 years and older with opioid use disorder (OUD) moderate or severe and who have not been taking prescribed medication for OUD (MOUD) for 14 days or more prior to hospitalization. Eligibility will be determined over one or more assessments during the index hospitalization. Once eligibility has been determined, participants will be randomized 1:1 to either a single injection of extended-release buprenorphine or TAU, which will include methadone, sublingual buprenorphine, or naltrexone. Connection to OUD care and ongoing MOUD following hospitalization will be per community standard. Participants will be assessed for engagement in OUD treatment by the presence of a legitimately prescribed MOUD on day 34 following hospital discharge. Further outcomes will be assessed at 90 and 180 days following hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized.
2. At least 18 years of age.
3. Meet Diagnostic and Statistical Manual (DSM-5) criteria for moderate or severe OUD.
4. Willing to initiate MOUD, including buprenorphine.
5. Able to speak English sufficiently to understand the study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

1. Anticipated length of stay less than 24-hours as determined by the ACS
2. Affected by a serious medical, psychiatric, or substance use disorder that, in the opinion of the study physician, would make it unsafe to participate in the study or may prevent collection of study data. This may include:

   1. Disabling terminal diagnosis for which discharge from hospital is not anticipated.
   2. Disabling terminal diagnosis for which hospice care is being sought.
   3. Severe alcohol or benzodiazepine use disorder that is anticipated to require complex medical detoxification which cannot be completed prior to randomization.
3. Taking a long-acting opioid other than buprenorphine (e.g., methadone, extended-release oxycodone, extended-release morphine) in the three consecutive days prior to randomization.
4. Liver enzyme tests (Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT)) more than 5 times upper limit of normal or chronic decompensated liver disease.
5. Currently pregnant.
6. Known allergy to buprenorphine or components of Atrigel delivery system.
7. Receipt of MOUD in the 14 days prior to hospitalization as maintenance treatment; however, patients may have received MOUD for withdrawal management during or prior to hospitalization at the time of enrollment.
8. Are currently in jail, prison or other overnight facility as required by court of law and/or is considered a prisoner under local law or is under current terms of civil commitment or guardianship.
9. Previously randomized as a participant in the study - individuals may only be enrolled and randomized once.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
The proportion of participants engaged in OUD care on the 34th day following hospital discharge. | 34 days post discharge from hospital
  Engagement in OUD is defined as coverage with a legitimately prescribed MOUD on that 34th day regardless of the source of prescribed MOUD coverage (e.g., formalized treatment program, primary care, jail, etc.).

SECONDARY OUTCOMES:
Proportion of participants that experience Adverse Events (AE) | 34 days
  34-days following hospital discharge
Proportion of participants engaged with MOUD | Days 90 and 180 post hospital discharge
  90- and 180-days following hospital discharge
Proportion of participants with positive urine drug test | Days 34, 90 and 180 post hospital discharge
  for illicit opioids 34-, and 90-, and 180-days following hospital discharge
Proportion of participants with self-reported opioid use | Days 34, 90 and 180 post hospital discharge
Self-reported 30- and 90-day hospital readmission rates | Days 30 and 90 post hospital discharge
Self-reported 30- and 90-day Emergency Department (ED) visit rates | Days 30 and 90 post hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Bart, MD,PhD, Principal Investigator — Hennepin Healthcare
Locations (6):
- United States (6):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - Hennepin Healthcare Research Institute, Minneapolis, Minnesota
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Data will be transmitted by the study Data and Statistics Center to the designated party for de-identification, posting, storing, and archiving on the National Institute on Drug Abuse (NIDA) Data Share website. Data Share is an online repository of data from studies funded by the National Institute on Drug Abuse. De-identified individual participant data is expected to be made available.
Supporting Information: Study Protocol
Time Frame: The data will be shared after the primary outcome paper has been accepted for publication, or 18 months after data lock, whichever comes first. The data will remain indefinitely.
Access Criteria: Data from this study will be available to researchers on the website https://datashare.nida.nih.gov/ after the study is complete and the data is analyzed. This website will not include information that can identify individual study participants.The following information will be posted: Study protocol, reference to study publication of primary outcome, data sets (SAS and ASCII ), annotated case report forms, define file (also known as Data Dictionary), study-specific de-identification notes. Prior to downloading any study data, the user will be prompted to complete a registration agreement for data use. Users will have to register a name and valid e-mail address in order to download data and to accept their responsibility for using data in accordance with the NIDA Data Share Agreement.
URL: https://datashare.nida.nih.gov/

REFERENCES:
- [Background] Liebschutz JM, Crooks D, Herman D, Anderson B, Tsui J, Meshesha LZ, Dossabhoy S, Stein M. Buprenorphine treatment for hospitalized, opioid-dependent patients: a randomized clinical trial. JAMA Intern Med. 2014 Aug;174(8):1369-76. doi: 10.1001/jamainternmed.2014.2556. PMID 25090173
- [Background] Lofwall MR, Walsh SL, Nunes EV, Bailey GL, Sigmon SC, Kampman KM, Frost M, Tiberg F, Linden M, Sheldon B, Oosman S, Peterson S, Chen M, Kim S. Weekly and Monthly Subcutaneous Buprenorphine Depot Formulations vs Daily Sublingual Buprenorphine With Naloxone for Treatment of Opioid Use Disorder: A Randomized Clinical Trial. JAMA Intern Med. 2018 Jun 1;178(6):764-773. doi: 10.1001/jamainternmed.2018.1052. PMID 29799968
- [Background] Trowbridge P, Weinstein ZM, Kerensky T, Roy P, Regan D, Samet JH, Walley AY. Addiction consultation services - Linking hospitalized patients to outpatient addiction treatment. J Subst Abuse Treat. 2017 Aug;79:1-5. doi: 10.1016/j.jsat.2017.05.007. Epub 2017 May 11. PMID 28673521
- [Derived] Bart G, Barth KS, Baukol P, Enns E, Ghitza UE, Harris J, Jelstrom E, Liebschutz JM, Magane KM, Voronca D, Weinstein ZM, Korthuis PT. Exemplar Hospital Initiation Trial to Enhance Treatment Engagement (EXHIT ENTRE): protocol for CTN-0098 an open-label randomized comparative effectiveness trial of extended-release buprenorphine versus treatment as usual on post-hospital treatment engagement for hospitalized patients with opioid use disorder. Addict Sci Clin Pract. 2024 Dec 2;19(1):91. doi: 10.1186/s13722-024-00510-5. PMID 39623502